CLINICAL TRIAL: NCT01141426
Title: Halifax Treatment Refractory Depression Trial: A Randomized Controlled Trial of Intensive Short-Term Dynamic Psychotherapy (ISTDP) Compared to Secondary Care Treatment as Usual
Brief Title: Halifax Treatment Refractory Depression Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joel Town (Other)
Collaborators: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Joel Town, Dr. Joel Town, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AA002
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Depression
Keywords: depression; treatment-resistance; psychodynamic psychotherapy; Treatment refractory depression
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secondary Care Treatment as Usual (Active Comparator): At the four secondary health care sites, treatment as usual will consist of a multidisciplinary team approach including pharmacotherapy and clinical management, supportive or structured activities focused around symptom management and in some cases, individual or group psychotherapy. Pharmacotherapy treatment strategies will be individualized regimes informed by evidence-based recommendations. TAU will not be regulated in order to get a naturalistic assessment of standard secondary care treatment delivery with the exception that trial participants not be offered a psychodynamic / psychoanalytic based psychotherapy treatment during the course of the trial. Therapeutic interventions are likely to be heterogeneous therefore the trial coordinator will document in detail the dose and approaches delivered to each participant in order to account for this heterogeneity.
  Interventions: Behavioral: Secondary Care Treatment as Usual
- Intensive Short-Term Dynamic Psychotherapy (ISTDP) Group (Experimental): The ISTDP model is an emotion focused brief format of psychotherapy that helps the patients identify and address emotional factors that culminate into exacerbation of depression and perpetuation of depression. The emphasis is on awareness of emotions and how they affect the person's behavioral patterns and mood. The research protocol calls for the treatment to be delivered according to a 20-session time-limited format. The first session is an extended 2-3 hour appointment (21), then sessions are planned to occur on a weekly basis lasting 60 minutes in duration. Termination in fewer sessions is based upon agreement between therapist and patient.
  Interventions: Behavioral: Intensive Short-term Dynamic Psychotherapy

INTERVENTIONS:
Behavioral: Intensive Short-term Dynamic Psychotherapy — The ISTDP model is an emotion focused brief format of psychotherapy that helps the patients identify and address emotional factors that culminate into exacerbation of depression and perpetuation of depression. The emphasis is on awareness of emotions and how they affect the person's behavioral patterns and mood. The research protocol calls for the treatment to be delivered according to a 20-session time-limited format. The first session is an extended 2-3 hour appointment (21), then sessions are planned to occur on a weekly basis lasting 60 minutes in duration. Termination in fewer sessions is based upon agreement between therapist and patient.
  Arms: Intensive Short-Term Dynamic Psychotherapy (ISTDP) Group
Behavioral: Secondary Care Treatment as Usual — At the four secondary health care sites, treatment as usual will consist of a multidisciplinary team approach including pharmacotherapy and clinical management, supportive or structured activities focused around symptom management and in some cases, individual or group psychotherapy. Pharmacotherapy treatment strategies will be individualized regimes informed by evidence-based recommendations. TAU will not be regulated in order to get a naturalistic assessment of standard secondary care treatment delivery with the exception that trial participants not be offered a psychodynamic / psychoanalytic based psychotherapy treatment during the course of the trial. Therapeutic interventions are likely to be heterogeneous therefore the trial coordinator will document in detail the dose and approaches delivered to each participant in order to account for this heterogeneity.
  Arms: Secondary Care Treatment as Usual

SUMMARY:
This study will use a randomized parallel group design to examine the effects of Intensive Short-term Dynamic Psychotherapy (ISTDP) for depressed patients non-remitting following at least one course of antidepressants. The effects of ISTDP will be judged through comparison against secondary care treatment as usual. The aim is to establish the clinical and cost effectiveness of ISTDP treatment.

DETAILED DESCRIPTION:
Major depression is a common morbid condition resulting in chronicity, recurrent disability, loss of physical health, and in many cases, death through suicide or medical conditions. By 2020, depression is projected to account for 4.4% of global disease burden (1) and the loss of 65 million disability-adjusted life years (2). A United Kingdom study (3) estimated direct treatment costs would reach three billion pounds by 2026 and indirect costs have been found to be 23 times larger (4).

Anti-depressant treatment is considered a bona fide first line agent for major depression. In some real-world studies, however, anti-depressant medications have not fared well. A large scale report, including the STAR-D study, reports remission rates that are disappointing: the percentage of patients attaining remission in first line and second line trials was 37% and 31% with relapse rates of 40% and 55%, respectively (5). Studies show that when depression does not remit with first line medication, it is more common to consider medication changes rather than commencing psychotherapy (6, 7). For treatment refractory depression (TRD), this situation may be due to insufficient empirical evidence demonstrating the efficacy of psychotherapy.

Current Canadian guidelines for depression (8) recommend psychodynamic psychotherapy as a third-line individual psychotherapy treatment option for major depressive disorder. However, two systematic reviews (9, 10) failed to identify any controlled trial data for any psychodynamic therapy for TRD and only three good quality randomized controlled trials (RCT) for other psychotherapy approaches. Although the empirical evidence for psychotherapy was described as limited, the authors concluded that it appears to be an effective option for TRD (10). Practitioners continue to provide psychodynamic therapies in routine clinical practice despite the shortage of empirical evidence; this suggests that formal study of psychodynamic therapies for TRD are urgently needed.

Within this broad treatment rubric, Short-Term Psychodynamic Psychotherapy (STPP) is a category of treatments derived from psychoanalytic theories but by definition distinguishable by the time-limited focus and emphasis on symptom reduction, in comparison to longer-term models where treatment is less structured and the therapist is typically less active. Interventions used in STPPs can be understood on a continuum between 'supportive' and 'expressive' techniques (11). More expressive therapies (e.g., ISTDP) emphasize greater attention to defences and anxiety that block the experiencing of underlying emotions. These emotional factors are understood to culminate in the exacerbation and perpetuation of depression. A meta-analysis found STPPs to be superior to control modalities in studies of major depression (Cohen's d = 0.69) but that further high-quality, randomized control trials are required (12). Of paramount importance however, the gains obtained with STPPs were maintained in long-term follow-up. Three studies have demonstrated direct treatment intervention outcome relationships between STPP and subsequent improvements in depressive symptoms (13-15).

One subtype of STPP is a method called Intensive Short Term Dynamic Psychotherapy (ISTDP). ISTDP has been studied in 18 published clinical studies. Randomized controlled trials have demonstrated its beneficial effects in patients with personality disorders, panic disorder and somatoform disorders (16-18). In a single case series of patients with treatment resistant depression, patients fared well with ISTDP with 8 of 10 achieving complete remission (19). These patients responded to a relatively short course of treatment with reduction and stoppage of the majority of medications. At the Centre for Emotions & Health (CEH), data were collected from a naturalistic sample of non-psychotic patients presenting with depression. The number of sessions varied from 2 to 62, with a mean (SD) of 8(11). Self-report scores on the Brief Symptom Inventory (BSI) (20) (N = 95) and Inventory of Interpersonal Problems (IIP) (21) (N = 84) were collected at time of intake and termination of ISTDP. The severity of clinical symptoms was markedly and significantly reduced after treatment.

Eight published studies have evaluated the cost-effectiveness of ISTDP (16, 19, 22-26). Two studies included patients with major depression. In one study of treatment-resistant depression (n = 10), we saw major drops in disability cost as 4 of 5 disabled patients returned to work and medications were stopped or reduced (19). In the second study of 231 patients with major depression now being analyzed (Abbass, in preparation), there was a $4,400 hospital and physician cost saving maintained year over year, while waiting list controls had no significant change over time. The post treatment cost savings in the subsequent 3 years were $5000, $5900 and $5100 per patient, thus supporting the concept of lasting cost reductions after treatment with ISTDP.

In summary, based on these preliminary empirical data highlighting the effectiveness of ISTDP, coupled with the current paucity of empirical support for all psychotherapies with this population, formal study of the efficacy of this approach for treatment refractory depression is warranted in the setting of a controlled efficacy trial. As a relatively brief and non-invasive treatment option, should research demonstrate evidence of cost effectiveness and clinical efficacy, this would support the call for this treatment to be made more readily available.

ELIGIBILITY:
Inclusion criteria:

* Patients aged 18 - 65 years.
* Patients must identify depression as their primary problem (rather than being secondary to other mental health diagnosis).
* Any DSM-IV diagnosis of Major Depression as assessed by the Mini Neuropsychiatric Interview plus (M.I.N.I. plus) at time of research intake interview.
* Patients will have had at least one treatment trial of antidepressants at an acceptable therapeutic dose (length ≥ 6 weeks) for the current depressive episode without adequate response (score on the Hamilton Rating Scale for Depression ≥ 16 ) at time of screening interview.
* Patients will not have started new medications in the previous ≥ 6 weeks, or have received psychotherapy treatment in the 12 months prior to being invited to participate in the study.
* Participants will agree to video-taped sessions and will consent to the investigator accessing their information in clinical files and hospital database (e.g., medications, number of visits to health care professionals).

Exclusion criteria

* Psychotic depression, bipolar depression, substance dependence, severe cluster A or B personality disorders, active suicidality, or cognitive impairment: such that patients require an intervention other than psychotherapy (as per the current protocol for the experimental treatment arm) or patients unable to give consent to treatment.
* Patients with depression due to a general medical condition or secondary to a comorbid mental health or psychosocial condition will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression | Baseline, 3, 6, 12, 18 months

SECONDARY OUTCOMES:
7-item Generalized Anxiety Disorder Scale (GAD-7) | Baseline, 3, 6, 9, 12, 18 months
Inventory of Interpersonal Problems 32-item | Baseline, 3, 6, 9, 12, 18 months
Toronto Alexithymia Scale | Baseline, 6, 9, 12, 18 months
12-item Short-Form Health Survey (SF-12) | Baseline, 3, 6, 12, 18 months
Clinical Outcomes in Routine Evaluation Outcome Measure (CORE-OM) | Baseline, 3, 6, 9, 12, 18 months
Trimbos and Institute of medical technology Assessment Cost Questionnaire for Psychiatry | Baseline, 6, 12, 18 months
9-item Patient Health Questionnaire (PHQ-9) | Baseline, 3, 6, 9, 12, 18 months
Patient Health Questionnaire-somatic symptom scale (PHQ-12) | Baseline, 3, 6, 9, 12, 18-month
Mini International Neuropsychiatric Inventory plus (M.I.N.I. plus) | Baseline, 6 months
Computerized Assessment SCID for DSM-IV (CAS-II) | Baseline, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel Town, Principal Investigator — Capital District Health Authority and Dalhousie University
Locations (1):
- Capital District Health Authority, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Guilbert JJ. The world health report 2002 - reducing risks, promoting healthy life. Educ Health (Abingdon). 2003 Jul;16(2):230. doi: 10.1080/1357628031000116808. No abstract available. PMID 14741909
- [Background] 2. Murray CJL, Lopez AD. The Global Burden of Disease. A Comprehensive Assessment of Mortality and Disability from Diseases, Injuries and Risk Factors in 1990 and Projected to 2020. Cambridge, Massachussetts: Harvard University Press; 1997.
- [Background] 3. McCrone P, Dhanasiri S, Patel A, Knapp M, Lawton-Smith S. Paying the Price: The Cost of Mental Health Care in England to 2026. London: King's Fund; 2008.
- [Background] Thomas CM, Morris S. Cost of depression among adults in England in 2000. Br J Psychiatry. 2003 Dec;183:514-9. doi: 10.1192/bjp.183.6.514. PMID 14645022
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Markowitz JC. When should psychotherapy be the treatment of choice for major depressive disorder? Curr Psychiatry Rep. 2008 Dec;10(6):452-7. doi: 10.1007/s11920-008-0073-7. PMID 18980727
- [Background] Simon GE, Ludman E, Unutzer J, Bauer MS. Design and implementation of a randomized trial evaluating systematic care for bipolar disorder. Bipolar Disord. 2002 Aug;4(4):226-36. doi: 10.1034/j.1399-5618.2002.01190.x. PMID 12190711
- [Background] Parikh SV, Segal ZV, Grigoriadis S, Ravindran AV, Kennedy SH, Lam RW, Patten SB; Canadian Network for Mood and Anxiety Treatments (CANMAT). Canadian Network for Mood and Anxiety Treatments (CANMAT) clinical guidelines for the management of major depressive disorder in adults. II. Psychotherapy alone or in combination with antidepressant medication. J Affect Disord. 2009 Oct;117 Suppl 1:S15-25. doi: 10.1016/j.jad.2009.06.042. Epub 2009 Aug 13. PMID 19682749
- [Background] Stimpson N, Agrawal N, Lewis G. Randomised controlled trials investigating pharmacological and psychological interventions for treatment-refractory depression. Systematic review. Br J Psychiatry. 2002 Oct;181:284-94. doi: 10.1192/bjp.181.4.284. PMID 12356654
- [Background] Trivedi RB, Nieuwsma JA, Williams JW Jr. Examination of the utility of psychotherapy for patients with treatment resistant depression: a systematic review. J Gen Intern Med. 2011 Jun;26(6):643-50. doi: 10.1007/s11606-010-1608-2. Epub 2010 Dec 24. PMID 21184287
- [Background] 11. Luborsky L. Principles of psychoanalytic psychotherapy: A manual for supportive/expressive treatment New York: Basic Books; 1984.
- [Background] Driessen E, Cuijpers P, de Maat SC, Abbass AA, de Jonghe F, Dekker JJ. The efficacy of short-term psychodynamic psychotherapy for depression: a meta-analysis. Clin Psychol Rev. 2010 Feb;30(1):25-36. doi: 10.1016/j.cpr.2009.08.010. PMID 19766369
- [Background] Barber JP, Crits-Christoph P, Luborsky L. Effects of therapist adherence and competence on patient outcome in brief dynamic therapy. J Consult Clin Psychol. 1996 Jun;64(3):619-22. doi: 10.1037//0022-006x.64.3.619. PMID 8698958
- [Background] 14. Gaston L, Thompson L, Gallagher D, Cournoyer L-G, Gagnon R. Alliance, technique, and their interactions in predicting outcome of behavioral, cognitive, and brief dynamic therapy. Psychotherapy Research. 1998;8(2):190-209.
- [Background] Hilsenroth MJ, Ackerman SJ, Blagys MD, Baity MR, Mooney MA. Short-term psychodynamic psychotherapy for depression: an examination of statistical, clinically significant, and technique-specific change. J Nerv Ment Dis. 2003 Jun;191(6):349-57. doi: 10.1097/01.NMD.0000071582.11781.67. PMID 12826915
- [Background] Abbass A, Sheldon A, Gyra J, Kalpin A. Intensive short-term dynamic psychotherapy for DSM-IV personality disorders: a randomized controlled trial. J Nerv Ment Dis. 2008 Mar;196(3):211-6. doi: 10.1097/NMD.0b013e3181662ff0. PMID 18340256
- [Background] Abbass A, Kisely S, Kroenke K. Short-term psychodynamic psychotherapy for somatic disorders. Systematic review and meta-analysis of clinical trials. Psychother Psychosom. 2009;78(5):265-74. doi: 10.1159/000228247. Epub 2009 Jul 11. PMID 19602915
- [Background] Abbass A, Town J, Driessen E. Intensive short-term dynamic psychotherapy: a systematic review and meta-analysis of outcome research. Harv Rev Psychiatry. 2012 Mar-Apr;20(2):97-108. doi: 10.3109/10673229.2012.677347. PMID 22512743
- [Background] Abbass AA. Intensive Short-Term Dynamic Psychotherapy of treatment-resistant depression: a pilot study. Depress Anxiety. 2006;23(7):449-52. doi: 10.1002/da.20203. PMID 16845654
- [Derived] Town JM, Falkenstrom F, Abbass A, Stride C. The anger-depression mechanism in dynamic therapy: Experiencing previously avoided anger positively predicts reduction in depression via working alliance and insight. J Couns Psychol. 2022 Apr;69(3):326-336. doi: 10.1037/cou0000581. Epub 2021 Sep 30. PMID 34591500